CLINICAL TRIAL: NCT06497374
Title: FcRn Antagonists (Efgartigimod) for Acute Neuromyelitis Optica Spectrum Disorders (NMOSD) Attack: a Phase 2, Randomized Controlled Trial.
Brief Title: FcRn Antagonists (Efgartigimod) for Acute NMOSD Attack
Acronym: FACT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240426
Record Dates: First submitted 2024-06-16; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder; NMO Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Efgartigimod+IVMP group (Experimental): Patients will receive efgartigimod alpha via intravenous infusion at a dose of 10 mg/kg, each infusion lasting approximately 2 hours, on Week 0, 1, 2 and 3. Efgartigimod should be administered no later than the second day after initiation of high-dose intravenous methylprednisolone therapy. This is delivered intravenously at a dosage of 1,000 mg/day for five consecutive days, which is then reduced to 500 mg/day for the next three days, followed by 240 mg/day for another three days, and then 120 mg/day for an additional three days. Subsequently, the treatment shifts to oral prednisone, starting with 60 mg daily for seven days, then decreasing to 50 mg daily for the next seven days, followed by 40 mg daily for another seven days. Afterward, the prednisone dosage is reduced by 5 mg every two weeks until it reaches 10 mg. After Week 4, Inebilizumab to prevent relapse will be introduced according to the indication.
  Interventions: Drug: Efgartigimod Alfa Injection; Drug: High-dose intravenous methylprednisolone
- IVMP group (Experimental): Patients will be treated with injectable methylprednisolone sodium succinate as described in Arm A. After Week 4, Inebilizumab to prevent relapse will be introduced according to the indication.
  Interventions: Drug: High-dose intravenous methylprednisolone
- Efgartigimod group (Other): Patients will be treated with efgartigimod alpha injection via intravenous infusion at a dosage of 10 mg/kg, with each session lasting approximately 2 hours, on Week 0, 1, 2 and 3. After Week 4, Inebilizumab to prevent relapse will be introduced according to the indication.
  Interventions: Drug: Efgartigimod Alfa Injection

INTERVENTIONS:
Drug: Efgartigimod Alfa Injection — Efgartigimod+IVMP; IVMP; Efgartigimod
  Arms: Efgartigimod group; Efgartigimod+IVMP group
Drug: High-dose intravenous methylprednisolone — Efgartigimod+IVMP; IVMP; Efgartigimod
  Arms: Efgartigimod+IVMP group; IVMP group

SUMMARY:
NMOSD is an autoimmune disease of the central nervous system that predominantly affects the spinal cord and optic nerves. The objectives of this study are to assess the efficacy and safety of FcRn antagonists (efgartigmod) for treatment of patients with neuromyelitis optica spectrum disorders during acute phase who are anti-aquaporin-4 (AQP4) antibody-positive. The potential of efgartigimod, an IgG1 Fc fragment that competes with IgG for FcRn binding, thereby lowering IgG levels, warrants further investigation as a treatment for acute neuromyelitis optica spectrum disorders attacks. This study aims to evaluate the therapeutic potential of efgartigmod in acute NMOSD attack.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ages 18 to 75.
2. Meet the 2015 International Panel of Experts (IPND) diagnostic criteria for neuromyelitis optica spectrum disorders.
3. Acute EDSS nadir of 2.5-7.5, and a change of at least 0.5 points from baseline due to an acute relapse event.
4. Confirmation of serum AQP4-IgG antibody positivity using the CBA assay.
5. Confirmation of an acute attack of neuromyelitis optica spectrum disorders either with an acute optic neuritis and/or acute myelitis, defined as a worsening in the patient's signs and symptoms of neurological/visual impairment, an increase in the EDSS score, and symptoms lasting more than 24 hours and occurring more than 1 month since the last attack. Combination of imaging and clinical evaluation will be used to assess relapse and rule out a pseudorelapse.
6. New lesions or enhanced lesions need to be found in MRI.
7. Subjects who were receiving immunosuppressive therapy prior to the screening period will be required to agree to discontinue immunosuppression.
8. Treatment is stable at least 3 months.

Exclusion Criteria:

1. Other core clinical symptoms besides optic neuritis and myelitis.
2. Severe neuromyelitis optica spectrum disorder attack, which in the judgment of the investigator is not appropriate for this study. Severe is defined as requiring assisted ventilation or likely to require assisted ventilation during the study based on the judgment of the investigator.
3. Subjects with total IgG levels ≤ 6 g/L at screening.
4. Subjects with a B-cell count ≤ 5% of the lower limit of normal at screening.
5. Received high-dose intravenous methylprednisolone within 4 weeks prior to the screening period.
6. Received intravenous immunoglobulin, plasma exchange, or immunoadsorption treatment within 4 weeks prior to the screening period.
7. Received a vaccination within the first 4 weeks of the screening period or planned during the study.
8. Using of a monoclonal antibody or investigational drug not mentioned above that has immunomodulatory effects within 3 months or 5 half-lives (whichever is longer) prior to the screening period.
9. Subject is known to be allergic to any component of the study drug or any other FcRn drug or contrast medium for enhanced MRI.
10. Subject is known to have contraindications to taking methylprednisolone (for subjects in A and B group).
11. Subjects with clinically significant active infections (including unresolved or inadequately treated infections, including active tuberculosis) as assessed by the investigator.
12. Subjects with positive screening tests for hepatitis B and C who have received live or live attenuated vaccine within 6 weeks prior to baseline.
13. Subjects is known unable to taken MRI.
14. Subjects is known to have other ophthalmic disease that affect vision as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-07-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Neurological Disability - Expanded Disability Scale Score | Acute nadir to week4
  The Kurtzke Expanded Disability Status Scale (EDSS) was developed to measure the disability status of subjects with demyelinating disease. It allows an objective quantification of the level of functioning that could be widely and reproducibly used by researchers and health care providers. The EDSS provides a total score on a scale that ranges from 0 to 10 where 0 is normal and 10 is deceased. Increasing disability is reflected in an increasing EDSS score.

SECONDARY OUTCOMES:
Change of FS score and MRC score at Week 12. | Baseline to week 12.
  To evaluate changes in neurologic outcomes in subjects with acute attacks in subjects with AQP4-IgG antibody-positive neuromyelitis optica spectrum disorders who are treated with efgartigimod + IVMP versus IVMP alone at Week 12.
  The Functional System (FS) was developed to measure the function of seven systems, including visual functions (score 0-6), brainstem functions (score 0-5), pyramical functions (score 0-6), cerebellar functions (score 0-5, X is the condition that pyramidal weakness (BMRC grade 3 or worse in limb strength) or sensory deficits interfere with cerebellar testing), sensory functions (score 0-6), bowel and bladder functions (score 0-6), cerebral functions (score 0-5). Increasing disability of different functional system is reflected in an increasing FS score.
  Muscle Power Assessment (MRC) was developed to assess the muscle power of limbs. A score of 0-5 was used to grade the power. Increasing disability of muscle power is reflected in an decreasing MRC score.
Change of EDSS score, FS score, and MRC score at Week 4 and 24. | Baseline to Week 4 and Week 24.
  To evaluate changes in neurologic outcomes in subjects with acute attacks in subjects with AQP4-IgG antibody-positive neuromyelitis optica spectrum disorders who are treated with efgartigimod + IVMP versus IVMP alone at Week 4 and Week 24. The EDSS score, FS score MRC score was described as in outcome 2.
Change of EQ-5D-5L score. | Baseline to Week 4, 12 and 24.
  To evaluate changes in quality of life in subjects at Week 4, 12, 24.
Change of high-contrast visual acuity in subjects with acute optic neuritis. | Baseline to Week 4, 12 and 24.
  To evaluate changes in vision outcomes (High contrast visual acuity ) in subjects with acute optic neuritis post-treatment at Week 4, 12, 24.
Change of OCT measurements in subjects with acute optic neuritis. | Baseline to Week 4, 12 and 24.
  To evaluate changes in vision outcomes (OCT measures) in subjects with acute optic neuritis post-treatment at Week 4, 12, 24.
The proportion of participants requiring rescue treatment during the study period. | Baseline to Week 24.
  To evaluate the proportion of subjects requiring rescue treatment during the study period.
The incidence of adverse events in the subjects during the study period. | Baseline to Week 24.
  To evaluate the safety and tolerability of efgartigimod +IVMP versus IVMP alone.
The vital signs, clinical laboratory indices, and electrocardiogram records of the subjects during the study period. | Baseline to Week 24.
  To evaluate the vital signs, clinical laboratory parameters and electrocardiograms during the study.

OTHER OUTCOMES:
Change of serum total IgG levels. | Baseline to Week 4, 12 and 24.
  To evaluate changes in serum levels of total IgG in participants post-treatment at Week 4, 12, 24.
Change of serum AQP4-IgG antibody levels. | Baseline to Week 4, 12 and 24.
  To evaluate changes in serum levels of AQP4-IgG antibodies in participants post-treatment at Week 4, 12, 24.
Change of serum GFAP and NfL. | Baseline to Week 4, 12 and 24.
  To evaluate changes in serum GFAP and NfL levels in participants after treatment at Week 4, 12 and 24.
Change of the size and extent of MRI lesions. | Baseline to Week 4, 12 and 24.
  To evaluate changes in spinal cord imaging in participants with acute myelitis following a course of efgartigimod + IVMP versus IVMP alone at Week 4, 12 and 24.